CLINICAL TRIAL: NCT01705080
Title: IntErnational Non-randomized, Single-arm, Long-term Follow-up Study of Patients With Uncontrolled HyperTensioN
Brief Title: IntErnational Long-term Follow-up Study of Patients With Uncontrolled HyperTensioN
Acronym: EnligHTN-II
Status: Terminated | Type: Observational
Why Stopped: Abbott made a decision to not further develop the RDN program.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 1201
Record Dates: First submitted 2012-09-19; First posted 2012-10-12 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Hypertension; Blood Pressure
Keywords: Renal Denervation; Renal artery; EnligHTN™ Renal Denervation System; Renal Artery Ablation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- A - EnligHTN for Severe Resistant HTN: * Office systolic Blood Pressure ≥160 mmHg
  * Subject is taking ≥3 anti-hypertensive medications (including 1 diuretic), or subject has documented drug intolerance to 2 or more of the 4 major classes of anti-hypertensives (ACE/ARB, Calcium Channel Blockers, Beta Blockers, or diuretic) and is unable to take 3 anti-hypertensive drugs.
  * Patient has an estimated GFR ≥45 mL/min per 1.73 m^2 using the Modification of Diet in Renal Disease (MDRD) formula
  Interventions: Device: EnligHTN
- B - EnligHTN for Resistant HTN: * Office systolic Blood Pressure ≥140 mmHg
  * Subject is taking ≥3 anti-hypertensive medications (including 1 diuretic), or subject has documented drug intolerance to 2 or more of the 4 major classes of anti-hypertensives (ACE/ARB, Calcium Channel Blockers, Beta Blockers, or diuretic) and is unable to take 3 anti-hypertensive drugs.
  * Patient has an estimated GFR ≥45 mL/min per 1.73 m^2 using the Modification of Diet in Renal Disease (MDRD) formula
  Interventions: Device: EnligHTN
- C - EnligHTN for Resistant HTN & CKD: * Office systolic Blood Pressure ≥140 mmHg
  * Subject is taking ≥3 anti-hypertensive medications (including 1 diuretic), or subject has documented drug intolerance to 2 or more of the 4 major classes of anti-hypertensives (ACE/ARB, Calcium Channel Blockers, Beta Blockers, or diuretic) and is unable to take 3 anti-hypertensive drugs.
  * Patient has an estimated ≥15 GFR <45 mL/min per 1.73 m^2 using the Modification of Diet in Renal Disease (MDRD) formula
  Interventions: Device: EnligHTN

INTERVENTIONS:
Device: EnligHTN — Renal artery ablation with EnligHTN system used for all groups

SUMMARY:
The purpose of this post market clinical investigation is to further evaluate the safety and performance of the EnligHTN™ Renal Denervation System in the treatment of patients with uncontrolled hypertension.

DETAILED DESCRIPTION:
This is a post market, prospective, multicenter, non-randomized, single arm study of the EnligHTN™ Renal Denervation System. Approximately 500 subjects with uncontrolled hypertension will undergo renal artery ablation at approximately 40 investigational sites located internationally and will be followed up to five years post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age at time of consent
* Subject must be able and willing to provide written informed consent
* Subject must be able and willing to comply with the required follow-up schedule
* Subject has office Systolic Blood Pressure ≥ 140 mmHg at confirmatory visit
* Subject has a daytime mean Systolic Ambulatory Blood Pressure > 135 mmHg within 90 days prior to procedure
* Subject has established hypertension (diagnosed ≥12 month prior to baseline) and is on a guideline based drug regimen at a stable and fully tolerated dose consisting of ≥ 3 anti-hypertensive medications (including 1 diuretic) or subject has a documented drug intolerance to 2 or more of the 4 major classes of anti-hypertensives (ACE/ARB, Calcium Channel Blockers, Beta Blockers, or diuretic) and is unable to take 3 anti-hypertensive drugs.

Exclusion Criteria:

* Subject has significant renovascular abnormalities such as renal artery stenosis > 30%
* Subject has undergone prior renal angioplasty, renal denervation, indwelling renal stents, and/or abdominal aortic stent grafts
* Subject has hemodynamically significant valvular heart disease as determined by study investigator
* Subject has a life expectancy less than 12 months, as determined by the Investigator
* Subject is participating in another clinical study which has the potential to impact their hypertension management (pharmaceutical/device/homeopathic)
* Subject is pregnant, nursing, or of childbearing potential and is not using adequate contraceptive methods
* Subject has active systemic infection
* Subject has renal arteries with diameter(s) < 4 mm in diameter
* Subject has an estimated GFR <15 mL/min per 1.73 m^2 using the MDRD formula
* Subject had a renal transplant or is awaiting a renal transplant
* Subject has blood clotting abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with uncontrolled hypertension
Sampling Method: Non-Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2013-01-17 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2019-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melvin Lobo, MBChB PhD, Principal Investigator — NIHR Barts Cardiovascular Biomedical Research Unit; Stephen Worthley, MB BS PhD, Principal Investigator — Royal Adelaide Hospital
Locations (33):
- Australia (4):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Prince Charles Hospital, Chermside
  - Royal Melbourne Hospital - City Campus, Parkville
  - Royal Perth Hospital, Perth
- France (5):
  - CHU de Besancon - Jean Minjoz, Besançon, Franche-Comte
  - Institute Cardio. Paris-Sud-Institut Jacques Cartier, Paris, Massy
  - Hopital de la Croix Rousse, Lyon
  - St-Etienne CHU, Saint-Etienne
  - Hopital Civil - Universitaires de Strasbourg, Strasbourg
- Germany (11):
  - Klinikum Coburg GmbH, Coburg, Bavaria
  - Klinikum Ingolstadt GmbH, Ingolstadt, Bavaria
  - Kerckhoff-Klinik gGmbH, Bad Nauheim, Hesse
  - Herz-und Diabetes Zentrum NRW, Bad Oeynhausen, North Rhine-Westphalia
  - Uni-Klinik Leipzig, Intervent. Angiologie, Leipzig, Saxony
  - Universitats-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen
  - Jüdisches Krankenhaus Berlin, Berlin
  - Universitatsklinikum Essen (AoR), Essen
  - Universitatsklinikum des Saarlandes, Homburg
  - Klinikum der Johannes-Gutenberg-Universitat, Mainz
  - Krankenhaus der Barmherzigen Bruder, Trier
- University of Athens, Ippocration Hospital, Athens, Greece
- Italy (3):
  - Fondazione Toscana Gabriele Monasterio CNR, Massa, Tuscany
  - Policlinico S.Orsola Malpighi, Bologna
  - Centro Cardiologico Monzino, Milan
- Netherlands (2):
  - Haga Ziekenhuis Locatie Leyenburg, The Hague
  - UMC Utrecht, Utrecht
- Dunedin Public Hospital, Dunedin, New Zealand
- Norway (2):
  - Haukeland Universitetssykehus, Bergen
  - St. Olavs University Hospital, Trondheim
- Hospital Universitario Donostia, San Sebastián, Basque, Spain
- Sahlgrenska University Hospital Gothenburg, Gothenburg, Sweden
- United Kingdom (2):
  - NIHR Barts Cardiovascular Biomedical Research Unit, London
  - Northern General Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 276 subjects who underwent renal artery ablation fell into the analysis population of three predefined arms at 33 investigational sites located throughout Europe and Australia. The enrollment began on January 2013 and the last subject was enrolled on 06 September, 2016. The patients last follow-up visit occurred on 27 November, 2019.
Pre-assignment Details: Among the 353 subjects who were screened initially, 66 subjects did not receive the renal artery ablation procedure, 11 subjects received procedure but did not satisfy the definition of any arm. The 11 subjects who received RND procedure were followed up for exploratory analysis and considered as "unassigned arm". Of these subjects, 5 subjects completed the study, 6 subjects were withdrawn prior to study completion. Hence they were excluded during the endpoint and safety analyses.
Groups:
- A - EnligHTN for Severe Resistant HTN: * Office systolic Blood Pressure ≥160 mmHg
  * Participant is taking ≥3 anti-hypertensive medications (including 1 diuretic), or participant has documented drug intolerance to 2 or more of the 4 major classes of anti-hypertensives (ACE/ARB, Calcium Channel Blockers, Beta Blockers, or diuretic) and is unable to take 3 anti-hypertensive drugs.
  * Participant has an estimated GFR ≥45 mL/min per 1.73 m^2 using the Modification of Diet in Renal Disease (MDRD) formula
  EnligHTN: Renal artery ablation with EnligHTN system used for all groups
- B - EnligHTN for Resistant HTN: * Office systolic Blood Pressure ≥140 mmHg
  * Participant is taking ≥3 anti-hypertensive medications (including 1 diuretic), or participant has documented drug intolerance to 2 or more of the 4 major classes of anti-hypertensives (ACE/ARB, Calcium Channel Blockers, Beta Blockers, or diuretic) and is unable to take 3 anti-hypertensive drugs.
  * Participant has an estimated GFR ≥45 mL/min per 1.73 m^2 using the Modification of Diet in Renal Disease (MDRD) formula
  EnligHTN: Renal artery ablation with EnligHTN system used for all groups
- C - EnligHTN for Resistant HTN & CKD: * Office systolic Blood Pressure ≥140 mmHg
  * Participant is taking ≥3 anti-hypertensive medications (including 1 diuretic), or participant has documented drug intolerance to 2 or more of the 4 major classes of anti-hypertensives (ACE/ARB, Calcium Channel Blockers, Beta Blockers, or diuretic) and is unable to take 3 anti-hypertensive drugs.
  * Participant has an estimated ≥15 GFR <45 mL/min per 1.73 m^2 using the Modification of Diet in Renal Disease (MDRD) formula
  EnligHTN: Renal artery ablation with EnligHTN system used for all groups
Period: Overall Study
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Started | 147 | 101 | 28
Renal Artery Ablation Procedure | 147 | 101 | 28
Discharge Following Renal Artery Ablation Procedure | 147 | 100 (Reason Not Completed: Withdrawal by Subject=1) | 28
Completed | 72 | 49 | 12
Not Completed | 75 | 52 | 16
Not completed — Missed visit | 10 | 4 | 1
Not completed — Death | 4 | 4 | 6
Not completed — Withdrawal by Subject | 61 | 44 | 9

BASELINE CHARACTERISTICS:
Population: Among the 353 subjects who were screened initially, 66 subjects did not receive the renal artery ablation procedure, 11 subjects received procedure but did not satisfy the definition of any arm. The 11 subjects who received RND procedure were followed up for exploratory analysis and considered as "unassigned arm". Of these subjects, 5 subjects completed the study, 6 subjects were withdrawn prior to study completion. Hence they were excluded during the endpoint and safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD | Total
Number analyzed (Participants) | 147 | 101 | 28 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (10.0) | 58.0 (11.8) | 68.5 (8.0) | 60.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 26 | 10 | 100
  Male | 83 | 75 | 18 | 176
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Office Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic | 180.4 (22.3) | 160.8 (17.5) | 177.3 (22.3) | 172.9 (22.6)
  Diastolic | 97.1 (16.3) | 91.2 (13.3) | 90.6 (13.2) | 94.3 (15.2)
24-hour ambulatory blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: The number of participants analyzed includes subjects who were available at that time of analysis
  mmHg
    Systolic: number analyzed (Participants) | 135 | 93 | 24 | 252
    Systolic | 159.0 (16.3) | 147.4 (12.3) | 161.8 (19.3) | 155.0 (16.3)
    Diastolic: number analyzed (Participants) | 135 | 93 | 24 | 252
    Diastolic | 88.9 (13.1) | 87.0 (14.4) | 82.9 (15.6) | 87.6 (13.9)

OUTCOME MEASURES:

1. Primary Outcome: Mean Reduction in Office Systolic Blood Pressure From Baseline to 6 Months
Description: Office blood pressure corresponds to the blood pressure measured by the doctor or the nurse/staff in the office or in the clinic during the participant visit. Office Blood Pressure measurements was recorded as the average Blood Pressure of three measurements. If there was a change in medication after the office Blood Pressure assessment was completed an additional set of office Blood Pressure measurements was performed.
Time Frame: Baseline to 6 months
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 142 | 96 | 27
mmHg
  Baseline | 179.9 (22.3) | 160.8 (17.9) | 177.1 (22.7)
  6 Months | 163.2 (25.1) | 147.9 (17.2) | 158.7 (21.9)
  Change from baseline to 6 months | -16.7 (26.7) | -12.9 (21.8) | -18.3 (25.8)

2. Secondary Outcome: Acute Safety: Percentage of Participants With Peri-procedural Events Within 30 Days Post-procedure
Description: The peri-procedural events occurring within 30 days post procedure were summarized as the percentage of the number of participants with peri-procedural events within 30 days post procedure compared to the number of participants at baseline for that population.
Time Frame: 30 days post procedure
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 147 | 101 | 28
Participants | 49 | 37 | 8

3. Secondary Outcome: Midterm Safety: Percentage of Participants With New Renal Artery Stenosis and/or Aneurysm at Ablation Site at 6 Months
Description: The new renal artery stenosis (>50%) and/or aneurysm at the site of ablation per Renal Artery Imaging (CT/MR) was summarized at each follow-up visit as the percentage of patients who have stenosis and/or aneurysm. Kaplan-meier analysis was performed on the time to the first new renal artery stenosis and/or aneurysm at the site of ablation, as appropriate.
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 147 | 101 | 28
Participants | 0 | 0 | 0

4. Secondary Outcome: Midterm Safety: Mean Change in eGFR (mL/Min/1.73m²) From Confirmatory Visit to 6 Months
Description: Renal function change based on eGFR was summarized by computing the change of the eGFR at each follow-up visit compared to baseline for each patient with data available in both time points and calculating the mean and standard deviation of the eGFR change at those intervals.
Time Frame: Confirmatory visit to 6 months
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 131 | 93 | 27
mL/min/1.73m^2
  Confirmatory visit | 80.2 (20.2) | 78.6 (17.6) | 35.3 (8.2)
  6 months | 79.5 (24.7) | 79.6 (19.6) | 41.3 (12.7)
  Change from confirmatory visit to 6 months | -0.7 (14.4) | 1.1 (13.5) | 5.9 (11.6)

5. Secondary Outcome: Long Term Safety: Percentage of Participants With New Renal Artery Stenosis and/or Aneurysm at Ablation Site at 2 Years
Description: The new renal artery stenosis (>50%) and/or aneurysm at the site of ablation per RenalArtery Imaging (CT/MR) was summarized at each follow-up visit as the percentage of patients who have stenosis and/or aneurysm. Kaplan-meier analysis was performed onthe time to the first new renal artery stenosis and/or aneurysm at the site of ablation, as appropriate.
Time Frame: 2 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 147 | 101 | 28
Participants | 2 | 2 | 0

6. Secondary Outcome: Long Term Safety: Percentage of Participants With New Renal Artery Stenosis and/or Aneurysm at Ablation Site at 5 Years
Description: as for outcome 5
Time Frame: 5 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 147 | 101 | 28
Participants | 3 | 2 | 0

7. Secondary Outcome: Long Term Safety: Mean Change in eGFR (mL/Min/1.73m²) From Confirmatory Visit to 2 Years
Description: as for outcome 4
Time Frame: Confirmatory visit to 2 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 103 | 81 | 20
mL/min/1.73m^2
  Confirmatory visit | 79.4 (17.4) | 78.4 (19.0) | 36.3 (8.2)
  2 years | 76.4 (21.6) | 77.7 (19.0) | 41.1 (14.1)
  Change from confirmatory visit to 2 years | -3.0 (15.8) | -0.7 (14.9) | 4.8 (13.2)

8. Secondary Outcome: Long Term Safety: Mean Change in eGFR (mL/Min/1.73m²) From Confirmatory Visit to 5 Years
Description: as for outcome 4
Time Frame: Confirmatory visit to 5 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 63 | 43 | 12
mL/min/1.73 m^2
  Confirmatory visit | 77.6 (14.7) | 80.8 (17.2) | 38.6 (7.5)
  5 years | 67.9 (20.0) | 77.0 (18.6) | 37.5 (16.5)
  Change from confirmatory visit to 5 years | -9.7 (17.3) | -3.8 (15.7) | -1.1 (14.5)

9. Secondary Outcome: Mean Change in Ambulatory Systolic Blood Pressure From Baseline to 6 Months
Description: 24-hour Ambulatory Blood Pressure measurements were taken according to Standard Joint National Committee VII Guidelines / ESC and ESH Guidelines at each follow-up visit. In the 24-hour blood pressure monitoring, the blood pressure of patient was measured every 30 minutes during the daytime and every 60 minutes during the night time. When using ABP, it was ensured that at least two measurements per hour are taken during the person's usual waking hours and 1 measurement per hour are taken during the person's usual night time hours. The average value of at least 14 measurements taken during the person's usual waking hours and average of at least 8 measurements taken during the person's usual sleeping hours were used for calculation of mean value.
Time Frame: Baseline to 6 months
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 121 | 85 | 21
mmHg
  Baseline | 158.3 (15.7) | 147.0 (12.1) | 160.4 (18.9)
  6 months | 151.2 (18.2) | 142.7 (17.3) | 152.2 (15.9)
  Change from baseline to 6 months | -7.1 (16.5) | -4.3 (17.1) | -8.1 (24.6)

10. Secondary Outcome: Mean Change in Ambulatory Diastolic Blood Pressure From Baseline to 6 Months
Description: as for outcome 9
Time Frame: Baseline to 6 months
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 121 | 85 | 21
mmHg
  Baseline | 88.8 (12.7) | 86.8 (14.3) | 83.3 (15.8)
  6 months | 85.5 (12.1) | 83.0 (12.5) | 78.1 (13.9)
  Change from baseline to 6 months | -3.3 (9.3) | -3.8 (13.4) | -5.1 (13.1)

11. Secondary Outcome: Mean Change in Office Diastolic Blood Pressure From Baseline to 6 Months
Description: as for outcome 1
Time Frame: Baseline to 6 months
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 142 | 96 | 27
mmHg
  Baseline | 97.0 (16.2) | 91.2 (13.6) | 91.0 (13.3)
  6 months | 89.6 (15.6) | 86.0 (13.4) | 77.9 (14.4)
  Change from baseline to 6 months | -7.4 (13.9) | -5.2 (12.2) | -13.1 (10.1)

12. Secondary Outcome: Percentage of Participants Achieved Office Systolic Blood Pressure < 140 mmHg at 6 Months
Description: The percentage of participants achieved office systolic blood pressure <140 mmHg at 6 months visit was computed as the percentage of the ratio of number of participants who achievied office systolic blood pressure <140 mmHg at 6 months visit to the number of participants with data available in 6 months visit.
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 142 | 96 | 27
Participants | 19 | 27 | 4

13. Secondary Outcome: Mean Change in Office Systolic Blood Pressure From Baseline to 1 Year Post Denervation
Description: as for outcome 1
Time Frame: Baseline to 1 year
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 132 | 94 | 26
mmHg
  Baseline | 180.0 (22.4) | 160.1 (17.6) | 176.8 (23.0)
  1 year | 166.4 (25.6) | 147.8 (20.8) | 159.8 (26.6)
  Change from baseline to 1 year | -13.6 (26.6) | -12.3 (22.6) | -17.0 (28.7)

14. Secondary Outcome: Mean Change in Office Systolic Blood Pressure From Baseline to 2 Years Post Denervation
Description: as for outcome 1
Time Frame: Baseline to 2 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 117 | 85 | 23
mmHg
  Baseline | 178.7 (22.0) | 158.5 (16.6) | 178.0 (22.4)
  2 years | 160.6 (26.5) | 144.3 (19.5) | 153.1 (17.5)
  Change from baseline to 2 years | -18.1 (29.0) | -14.2 (20.9) | -24.8 (27.0)

15. Secondary Outcome: Mean Change in Office Systolic Blood Pressure From Baseline to 3 Years Post Denervation
Description: as for outcome 1
Time Frame: Baseline to 3 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 97 | 72 | 20
mmHg
  Baseline | 179.3 (21.9) | 160.7 (17.5) | 179.0 (23.7)
  3 years | 159.1 (28.5) | 143.8 (19.4) | 151.2 (21.3)
  Change from baseline to 3 years | -20.2 (34.1) | -16.9 (23.1) | -27.8 (28.1)

16. Secondary Outcome: Mean Change in Office Systolic Blood Pressure From Baseline to 4 Years Post Denervation
Description: as for outcome 1
Time Frame: Baseline to 4 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 90 | 68 | 18
mmHg
  Baseline | 177.7 (21.8) | 157.6 (15.4) | 180.4 (24.1)
  4 years | 156.2 (28.8) | 144.6 (25.3) | 146.9 (23.5)
  Change from baseline to 4 years | -21.5 (35.4) | -13.0 (24.9) | -33.5 (24.4)

17. Secondary Outcome: Mean Change in Office Systolic Blood Pressure From Baseline to 5 Years Post Denervation
Description: as for outcome 1
Time Frame: Baseline to 5 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 71 | 49 | 12
mmHg
  Baseline | 176.2 (20.3) | 160.2 (16.3) | 184.8 (24.6)
  5 years | 151.8 (22.6) | 144.4 (21.8) | 152.8 (19.1)
  Change from baseline to 5 years | -24.4 (28.4) | -15.7 (24.8) | -32.0 (25.7)

18. Secondary Outcome: Mean Change in Office Diastolic Blood Pressure From Baseline to 1 Year Post Denervation
Description: as for outcome 1
Time Frame: Baseline to 1 year
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 132 | 94 | 26
mmHg
  Baseline | 97.8 (16.6) | 91.0 (13.5) | 91.5 (13.3)
  1 year | 90.9 (17.6) | 85.5 (13.7) | 78.5 (14.2)
  Change from baseline to 1 year | -6.9 (15.0) | -5.5 (13.2) | -13.0 (13.3)

19. Secondary Outcome: Mean Change in Office Diastolic Blood Pressure From Baseline to 2 Years Post Denervation
Description: as for outcome 1
Time Frame: Baseline to 2 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 117 | 85 | 23
mmHg
  Baseline | 97.1 (16.8) | 91.0 (12.7) | 92.0 (12.9)
  2 years | 88.2 (16.6) | 83.4 (13.0) | 75.2 (14.3)
  Change from baseline to 2 years | -8.9 (16.5) | -7.6 (12.3) | -16.8 (14.7)

20. Secondary Outcome: Mean Change in Office Diastolic Blood Pressure From Baseline to 3 Years Post Denervation
Description: as for outcome 1
Time Frame: Baseline to 3 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 97 | 72 | 20
mmHg
  Baseline | 98.6 (17.5) | 92.0 (13.2) | 91.3 (13.3)
  3 years | 87.1 (15.8) | 82.9 (12.8) | 76.6 (14.8)
  Change from baseline to 3 years | -11.5 (18.4) | -9.0 (12.6) | -14.7 (14.5)

21. Secondary Outcome: Mean Change in Office Diastolic Blood Pressure From Baseline to 4 Years Post Denervation
Description: as for outcome 1
Time Frame: Baseline to 4 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 90 | 68 | 18
mmHg
  Baseline | 97.5 (17.5) | 91.0 (12.7) | 93.2 (11.2)
  4 years | 86.2 (13.5) | 85.2 (16.3) | 77.2 (12.3)
  Change from baseline to 4 years | -11.3 (18.2) | -5.9 (13.4) | -16.0 (9.8)

22. Secondary Outcome: Mean Change in Office Diastolic Blood Pressure From Baseline to 5 Years Post Denervation
Description: as for outcome 1
Time Frame: Baseline to 5 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 71 | 49 | 12
mmHg
  Baseline | 98.4 (17.3) | 93.1 (12.8) | 95.8 (13.0)
  5 years | 84.9 (11.7) | 85.1 (16.1) | 78.7 (12.7)
  Change from baseline to 5 years | -13.4 (14.4) | -8.0 (14.5) | -17.1 (14.0)

23. Secondary Outcome: Mean Change in Ambulatory Systolic Blood Pressure From Baseline to 1 Year Post Denervation
Description: as for outcome 9
Time Frame: Baseline to 1 year
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 105 | 78 | 19
mmHg
  Baseline | 159.1 (16.1) | 146.8 (11.4) | 163.9 (18.8)
  1 year | 149.0 (18.7) | 141.7 (17.3) | 148.2 (21.1)
  Change from baseline to 1 year | -10.1 (18.3) | -5.1 (16.8) | -15.8 (24.3)

24. Secondary Outcome: Mean Change in Ambulatory Systolic Blood Pressure From Baseline to 2 Years Post Denervation
Description: as for outcome 9
Time Frame: Baseline to 2 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 92 | 70 | 16
mmHg
  Baseline | 158.5 (15.8) | 146.7 (11.8) | 159.9 (16.8)
  2 years | 148.0 (17.2) | 139.5 (15.0) | 144.0 (16.7)
  Change from baseline to 2 years | -10.5 (18.6) | -7.2 (16.0) | -15.9 (18.7)

25. Secondary Outcome: Mean Change in Ambulatory Systolic Blood Pressure From Baseline to 3 Years Post Denervation
Description: as for outcome 9
Time Frame: Baseline to 3 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 72 | 57 | 11
mmHg
  Baseline | 157.8 (15.9) | 147.0 (11.9) | 156.0 (14.8)
  3 years | 144.2 (19.3) | 139.8 (18.1) | 151.2 (18.8)
  Change from baseline to 3 years | -13.6 (21.5) | -7.2 (18.8) | -4.8 (20.5)

26. Secondary Outcome: Mean Change in Ambulatory Systolic Blood Pressure From Baseline to 4 Years Post Denervation
Description: as for outcome 9
Time Frame: Baseline to 4 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 67 | 56 | 12
mmHg
  Baseline | 157.2 (14.5) | 146.3 (11.7) | 158.4 (16.4)
  4 years | 142.3 (19.6) | 137.9 (19.1) | 151.6 (21.2)
  Change from baseline to 4 years | -14.9 (22.4) | -8.5 (17.8) | -6.8 (29.6)

27. Secondary Outcome: Mean Change in Ambulatory Systolic Blood Pressure From Baseline to 5 Years Post Denervation
Description: as for outcome 9
Time Frame: Baseline to 5 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 50 | 35 | 10
mmHg
  Baseline | 155.2 (14.9) | 143.7 (9.8) | 158.0 (18.1)
  5 years | 140.0 (17.8) | 133.3 (13.4) | 146.3 (26.3)
  Change from baseline to 5 years | -15.1 (22.0) | -10.4 (11.8) | -11.7 (33.4)

28. Secondary Outcome: Mean Change in Ambulatory Diastolic Blood Pressure From Baseline to 1 Year Post Denervation
Description: as for outcome 9
Time Frame: Baseline to 1 year
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 105 | 78 | 19
mmHg
  Baseline | 89.1 (12.9) | 86.2 (14.1) | 85.4 (16.3)
  1 year | 84.7 (12.0) | 81.9 (12.2) | 77.7 (12.2)
  Change from baseline to 1 year | -4.4 (10.4) | -4.4 (13.4) | -7.6 (14.1)

29. Secondary Outcome: Mean Change in Ambulatory Diastolic Blood Pressure From Baseline to 2 Years Post Denervation
Description: as for outcome 9
Time Frame: Baseline to 2 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 92 | 70 | 16
mmHg
  Baseline | 88.6 (13.2) | 86.6 (14.2) | 84.6 (16.9)
  2 years | 83.8 (12.0) | 81.5 (11.4) | 76.9 (14.8)
  Change from baseline to 2 years | -4.8 (10.4) | -5.0 (12.3) | -7.6 (10.8)

30. Secondary Outcome: Mean Change in Ambulatory Diastolic Blood Pressure From Baseline to 3 Years Post Denervation
Description: as for outcome 9
Time Frame: Baseline to 3 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 72 | 57 | 11
mmHg
  Baseline | 89.0 (12.9) | 87.7 (14.7) | 81.7 (14.7)
  3 years | 81.3 (11.2) | 81.2 (12.9) | 76.8 (12.9)
  Change from baseline to 3 years | -7.7 (13.8) | -6.5 (13.9) | -4.9 (10.5)

31. Secondary Outcome: Mean Change in Ambulatory Diastolic Blood Pressure From Baseline to 4 Years Post Denervation
Description: as for outcome 9
Time Frame: Baseline to 4 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 67 | 56 | 12
mmHg
  Baseline | 88.4 (12.5) | 87.6 (14.8) | 82.1 (14.1)
  4 years | 80.3 (12.5) | 80.9 (13.4) | 78.1 (12.6)
  Change from baseline to 4 years | -8.1 (14.6) | -6.6 (14.5) | -4.0 (11.6)

32. Secondary Outcome: Mean Change in Ambulatory Diastolic Blood Pressure From Baseline to 5 Years Post Denervation
Description: as for outcome 9
Time Frame: Baseline to 5 years
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
Number analyzed (Participants) | 50 | 35 | 10
mmHg
  Baseline | 87.1 (13.1) | 87.9 (15.6) | 83.2 (14.8)
  5 years | 79.2 (10.7) | 78.5 (11.1) | 76.0 (14.4)
  Change from baseline to 5 years | -7.8 (12.6) | -9.4 (13.1) | -7.2 (13.1)

ADVERSE EVENTS:
Time Frame: 5 years
Description: Among the 353 subjects who were screened initially, 66 subjects did not receive the renal artery ablation procedure, 11 subjects received procedure but did not satisfy the definition of any arm. The 11 subjects who received RND procedure were followed up for exploratory analysis and considered as "unassigned arm". Of these subjects, 5 subjects completed the study, 6 subjects were withdrawn prior to study completion. Hence they were excluded during the endpoint and safety analyses.
Arm/Group | A - EnligHTN for Severe Resistant HTN | B - EnligHTN for Resistant HTN | C - EnligHTN for Resistant HTN & CKD
All-Cause Mortality (participants affected / at risk) | 4/147 | 4/101 | 6/28
Serious Adverse Events (participants affected / at risk) | 72/147 | 38/101 | 18/28
Other Adverse Events (participants affected / at risk) | 40/147 | 26/101 | 9/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A - EnligHTN for Severe Resistant HTN (N=147) | B - EnligHTN for Resistant HTN (N=101) | C - EnligHTN for Resistant HTN & CKD (N=28)
Anemias (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Bleeding (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Trauma (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (6) | 1 (1) | 0 (0)
Anterior Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic Valve Stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 3 (3) | 3 (4) | 2 (2)
Atrial Flutter (Cardiac disorders) | 1 (1) | 1 (3) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid Aneurysm-Aneurysm Of Left Internal Carotid Artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 7 (7) | 4 (4) | 2 (2)
Congestive Heart Failure (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Decompensated Heart Failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
First Degree Heart/AV Block/Cardiac Arrhythmia - 1st degree AV Block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Heart Failure (Cardiac disorders) | 4 (5) | 2 (2) | 3 (4)
Myocardial Infarction (Cardiac disorders) | 5 (8) | 5 (5) | 3 (3)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Paroxysmal Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Persistent Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Right Ventricular Failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ST Segment Changes (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
SVC Syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Second Degree Heart Block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus Bradycardia/Sinus Bradycardia (Cardiac Arrhythmia) (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Unstable Angina (Cardiac disorders) | 5 (7) | 4 (6) | 1 (1)
Hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal Tear (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Perforated Appendix (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (General disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 1 (2) | 0 (0) | 0 (0)
Lacerations (General disorders) | 1 (1) | 0 (0) | 0 (0)
Melena (General disorders) | 0 (0) | 0 (0) | 1 (1)
Other-Bladder (General disorders) | 1 (1) | 0 (0) | 0 (0)
Other-Death (General disorders) | 0 (0) | 1 (1) | 1 (1)
Other-Death Of Unknown Cause (General disorders) | 0 (0) | 0 (0) | 1 (1)
Other-Hemorrhagic Lymphocele (General disorders) | 0 (0) | 0 (0) | 1 (1)
Other-Non-Specifc Acute Lung Injury (General disorders) | 0 (0) | 0 (0) | 1 (1)
Shock (General disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (General disorders) | 2 (2) | 2 (3) | 1 (1)
Vertigo (General disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Pancreatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial Infections (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial Infections of the Skin (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Chlamydial Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected Cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
Pneumonia in the Compromised Host (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Allergic Dye Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
In-Stent Restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Ankle Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Calf Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tendon Tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Benign Prostatic Hyperplasia (BPH) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Kidney Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Chronic Subdural Hematoma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis/Weakness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhagic Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Ischemic Stroke (Nervous system disorders) | 4 (4) | 2 (2) | 1 (1)
Lumbar Spondylosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure/Convulsions/Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Stroke (Nervous system disorders) | 7 (9) | 3 (3) | 0 (0)
Transient Ischemic Attack (TIA) (Nervous system disorders) | 6 (6) | 0 (0) | 0 (0)
Acute Renal Failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Chronic Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Kidney Pain/Flank Pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal Congestion-Urinary Obstruction-Renal Congestion (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Ureteral Dysfunction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urethral Dysfunction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infections (Renal and urinary disorders) | 1 (2) | 2 (2) | 0 (0)
Acute Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Common Cold/Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Mediastinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2)
Cutaneous Abcesses (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arterial Hypertension/Hypertension (Vascular disorders) | 10 (12) | 5 (7) | 2 (2)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral Arterial Occlusion (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Renal Artery Dissection (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Renal Artery Stenosis (Vascular disorders) | 6 (6) | 3 (4) | 0 (0)
Renovascular Hypertension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Thrombus (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
VASC Bleeding (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
VASC Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
VASC Pseudoaneurysm (Vascular disorders) | 1 (1) | 3 (3) | 0 (0)
Vasospasm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A - EnligHTN for Severe Resistant HTN (N=147) | B - EnligHTN for Resistant HTN (N=101) | C - EnligHTN for Resistant HTN & CKD (N=28)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Heart Failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mobitz II Block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sick Sinus Syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus Bradycardia/Sinus Bradycardia (Cardiac Arrhythmia) (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Eye Bleed (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colon Polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 1 (1) | 0 (0)
Edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Elective Procedure (General disorders) | 1 (1) | 1 (1) | 0 (0)
Elective Surgery (General disorders) | 3 (4) | 2 (2) | 0 (0)
Headache (General disorders) | 2 (2) | 0 (0) | 0 (0)
Numbness-Numbness In Right Thigh (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Other-Small Wedge Shaped Abnormalities In Both Kidneys In Keeping With Small Infarcts (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hip Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Low Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Muscle Twitch (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis/Degenerative Joint Disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Benign Mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Numbness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient Ischemic Attack (TIA) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Device Malposition or Malfunction (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Abnormal Renal Function (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Kidney Pain/Flank Pain (Renal and urinary disorders) | 5 (5) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Prostate Disease (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic Dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Artery Stenosis (Vascular disorders) | 7 (8) | 2 (2) | 0 (0)
VASC Bleeding (Vascular disorders) | 4 (4) | 2 (2) | 1 (1)
VASC Bruise (Vascular disorders) | 3 (3) | 2 (2) | 2 (2)
VASC Drainage (Vascular disorders) | 9 (9) | 3 (3) | 0 (0)
VASC Hematoma (Vascular disorders) | 5 (5) | 5 (5) | 1 (1)
VASC Pain (Vascular disorders) | 7 (7) | 5 (6) | 1 (1)
VASC Pseudoaneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
VASC Vessel Perforation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vaso Vagal Response (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vasospasm (Vascular disorders) | 15 (17) | 12 (17) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2012-11-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT01705080/Prot_SAP_ICF_000.pdf